CLINICAL TRIAL: NCT02837289
Title: Activation of Hip Muscles in Runners With Patellofemoral Syndrome: Double-blind Randomized Clinical Trial
Brief Title: Activation of Hip Muscles in Runners With Patellofemoral Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Christiane Macedo, first investigator, Universidade Estadual de Londrina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: therapy taping in runners
Record Dates: First submitted 2016-07-12; First posted 2016-07-19 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: patellofemoral pain syndrome; therapy taping; knee; physical therapy; runners
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Other): Therapy taping follows an anatomical pattern from the femur until tibia for correction of dynamic valgus with therapy taping.
  Interventions: Other: Therapy taping
- Placebo (Other): Placebo taping follows a different anatomical path without tension, eliminating all therapeutic process elements
  Interventions: Other: Placebo taping

INTERVENTIONS:
Other: Therapy taping — Therapy taping follows an anatomical pattern from the femur until tibia for correction of dynamic valgus with therapy taping.
  Arms: Treatment
Other: Placebo taping — Placebo taping follows a different anatomical path without tension, eliminating all therapeutic process elements
  Arms: Placebo

SUMMARY:
Introduction: Hip motor control deficit and neuromuscular disorders of the gluteus medius influence the mechanics of patellofemoral joints through increased dynamic knee valgus and can lead to Patellofemoral Pain Syndrome (PFPS). Mechanoreceptors can be stimulated by an elastic tape, which sends desired tactile cues via afferent improving the functional support of the musculoskeletal system.

Objective: To analyze the response to hip stabilizer muscle activation in street runners with PFPS through the application of elastic tape therapy.

Methods: The investigators evaluated street runners between the ages of 18 and 45, who run at least 5km/week and had been suffering from pain for at least 3 months. The volunteers had been assessed in relation to their measurements, experience of pain and training routine, their medius muscle (GM) and biceps femoris muscle (BF) had also been tested with surface electromyography through pre-determined performance tests. The participants of both groups wore a bandage for 6 weeks (1 per week). However for the participants of the placebo group the investigators applied a different anatomical path without tension, eliminating all the therapeutic elements. The volunteers were reassessed following the trial.

Hypothesis: Expected to observe that elastic tape therapy do result in any improvement in the activation of hip muscles and improvement of pain in street runners with patellofemoral pain syndrome.

DETAILED DESCRIPTION:
Will be recruited individuals 18-45 years of age, of at least running frequency 5 km/week and history of pain in the knee for at least three months in two or more of the following listed activities: up or down stairs, squatting, kneeling , jump, long time sitting or pain on palpation of the lateral side / medial patella.

Will be included individuals without cardiovascular diseases, which have not undergone surgery of the lower limbs in the last two years without back pain and without injury to the hip or knee. They will be excluded from those presenting allergy to the use of elastic bandage or who can not remain with the use of it during the stipulated period. Participants will sign an informed consent and informed, prior to the start of collections.

Data collection was developed with a electromyography (EMG) for muscle data and questionnaire with participants by a blinded examiner initially will be held. The questionnaire consists of the Visual Analogue Scale (VAS). For EMG of the gluteus medius (GM) and biceps femoris (BF), the electrodes are positioned according to the protocols of Surface Electromyography for the Non-Invasive Assessment of Muscles (SENIAM), with the reference electrode located in anterior tibial tuberosity. The application site will be prepared with abrasion and cleansing the skin with 70% alcohol and trichotomy. The maneuver of maximum voluntary isometric contraction (MVIC) will be trained and previously performed the collection, with five seconds support for normalization of data to the gluteus medius and biceps. Among the MVICs every muscle will hold a minute's rest. The muscle activity recorded during the exercises will be expressed in percentage of MVIC. After maneuvers MVIC, individuals will rest for five minutes and then immediately to start the acquisition of electromyographic data during functional tests.

For this, individuals previously will be guided and trained to realize them. During testing, barefoot athletes will be positioned on one foot on the leg with more intense pain complaints, contralateral leg approximately 70 ° of knee flexion, relaxed upper body next to the body, torso upright and keeping focused look a marking affixed to the wall at eye level. In the first test, prompted a squat (AG) of approximately 45 ° of knee flexion, with one foot; in the second test, the same squat will be held, but followed by maximum external rotation (ROT-AG) in the hip support. The cadence of the movement will be standardized and guided by the appraiser to be started and completed in 10 seconds. Functional tests are designed to simulate the action of the hip muscles in the race support phase and motor control of the lower limb.

After electromyographic reviews, be held to randomization to the control group and treatment through and opaque sealed envelopes, by a blinded evaluator. Individuals of both groups will be submitted to the application of the bandage on the leg with pain complaints. For this, a qualified professional trained for the bandage application in relation to anatomical landmarks and elastic tension of the application, without the knowledge, so as to physiology or function thereof. Will be used two techniques in the intervention group. For the placebo group, the application of the bandage will follow a different anatomical path without tension, eliminating all therapeutic process elements.

The groups will be followed for six weeks and will be guided them to keep their daily routine. Each week, individuals remain five days with the application of the bandage, and two days without, to avoid possible adverse effects of excessive and constant use of it. After this, a new bandage will be applied by the same trained professional, following the protocols already mentioned. After six weeks, the volunteers return for reevaluation.

ELIGIBILITY:
Inclusion Criteria: Clinical diagnosis of patellofemoral dysfunction issued by a specialist orthopedic knee and provide anterior knee pain of 3 or more on the Visual Analogue Scale (VAS) for a minimum of 8 weeks prior to evaluation;

* Previous retropatellar pain or knee, for at least 3 of the following: up / down stairs, squatting, running, kneeling, sitting for long periods and insidious onset of symptoms unrelated to trauma.

Exclusion Criteria:

* History of severe / traumatic knee injury, surgery history in the locomotor system;
* Patellar luxation history; clinical evidence of meniscus injury; ligamentous instability; patellar tendinitis.
* Presence of neurological, cardiovascular or rheumatologic diseases; pregnancy; diabetes,
* Abnormal sensitivity in the plantar;
* Medication and / or therapy in the last six months and hypersensitivity or allergy to tape.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-07-01; Primary Completion 2016-07-02 (Actual); Study Completion 2017-05-03 (Actual)

PRIMARY OUTCOMES:
Changes in muscle activation by electromyography after treatment with therapy taping | before and after 6 weeks of intervention
  Willy et al (2013) suggest that interventions that seek biomechanical correction of the hip can reduce retropatellar pressure and improve the pain and function of individuals with PFD. Thus, it is sought to increase or reduce muscular activation, with a response in the locomotor system, which is confirmed by Hsu (2009) evidencing the relation of the elastic bandage to the muscular activation level. Slupik et al (2007) sought to determine the effect of the elastic bandage on the medial vastus muscle tone during isometric contractions, and they concluded that the bandage offered better support for the musculoskeletal system.

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Macedo, doctor, Principal Investigator — Universidade Estadual de Londrina
Locations (1):
- university hospital of the State University of Londrina, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fukuda TY, Rossetto FM, Magalhaes E, Bryk FF, Lucareli PR, de Almeida Aparecida Carvalho N. Short-term effects of hip abductors and lateral rotators strengthening in females with patellofemoral pain syndrome: a randomized controlled clinical trial. J Orthop Sports Phys Ther. 2010 Nov;40(11):736-42. doi: 10.2519/jospt.2010.3246. PMID 21041965
- [Background] Willy RW, Davis IS. Varied response to mirror gait retraining of gluteus medius control, hip kinematics, pain, and function in 2 female runners with patellofemoral pain. J Orthop Sports Phys Ther. 2013 Dec;43(12):864-74. doi: 10.2519/jospt.2013.4516. Epub 2013 Oct 30. PMID 24175611
- [Background] Hsu YH, Chen WY, Lin HC, Wang WT, Shih YF. The effects of taping on scapular kinematics and muscle performance in baseball players with shoulder impingement syndrome. J Electromyogr Kinesiol. 2009 Dec;19(6):1092-9. doi: 10.1016/j.jelekin.2008.11.003. Epub 2009 Jan 14. PMID 19147374
- [Background] Slupik A, Dwornik M, Bialoszewski D, Zych E. Effect of Kinesio Taping on bioelectrical activity of vastus medialis muscle. Preliminary report. Ortop Traumatol Rehabil. 2007 Nov-Dec;9(6):644-51. English, Polish. PMID 18227756
- [Result] Thelen MD, Dauber JA, Stoneman PD. The clinical efficacy of kinesio tape for shoulder pain: a randomized, double-blinded, clinical trial. J Orthop Sports Phys Ther. 2008 Jul;38(7):389-95. doi: 10.2519/jospt.2008.2791. Epub 2008 May 29. PMID 18591761